CLINICAL TRIAL: NCT04280926
Title: Use of High Sensitivity Cardiac Troponin in Safely Ruling Out Emergency Patients with Acute Myocardial Injury and Infarction (SAFETY)
Brief Title: Use of High Sensitivity Cardiac Troponin in Ruling Out Emergency Patients with Acute Myocardial Injury and Infarction
Acronym: SAFETY
Status: Completed | Type: Observational
Sponsor: Hennepin Healthcare Research Institute (Other)
Collaborators: Siemens Healthineers (Unknown)
Responsible Party: Sponsor
Other Study IDs: SAFETY
Record Dates: First submitted 2020-01-23; First posted 2020-02-21 (Actual); Last update posted 2024-12-17 (Actual); Status verified 2024-10

CONDITIONS: Acute Myocardial Infarction; Acute Coronary Syndrome
Keywords: Troponin; high-sensitivity cardiac troponin; acute myocardial infarction; Siemens Atellica
MeSH Terms: conditions — Acute Coronary Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Excess blood is biobanked after clinical testing for cTnI
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Cohort: Study population: Prospective, observational cohort study of consecutives patients (goal, 2000 patients over 4 months) presenting to the emergency department, in whom serial cTnI measurements are ordered on clinical indication at Hennepin Healthcare / Hennepin County Medical Center (Minneapolis, MN, USA) to rule-in and rule-out acute myocardial infarction.
  Interventions: Diagnostic Test: Cardiac Troponin Testing

INTERVENTIONS:
Diagnostic Test: Cardiac Troponin Testing — Fresh serum or lithium heparin plasma samples will be measured with the Atellica IM TnIH assay (Siemens Heatlhineers).

SUMMARY:
Examine the analytical and clinical performance of Atellica IM TnIH assay for the diagnosis and rule out of acute myocardial injury and myocardial infarction in patients presenting to the emergency department in whom serial cTnI measurements are obtained on clinical indication.

DETAILED DESCRIPTION:
Background: Studies addressing the clinical performance of the Siemens Healthineers High-Sensitivity Troponin I assay (TnIH) on the Atellica IM analyzer for the diagnosis and rule out of acute myocardial injury and myocardial infarction in consecutive patients presenting to a United States (US) emergency department are lacking.

Study objective: Examine the analytical and clinical performance of Atellica IM TnIH assay for the diagnosis and rule out of acute myocardial injury and myocardial infarction in patients presenting to the emergency department in whom serial cTnI measurements are obtained on clinical indication.

Hypothesis: The Atellica IM TnIH assay will offer an excellent diagnostic performance for acute myocardial injury and acute myocardial infarction, as well as expedite the risk stratification of patients for early discharge from the emergency department.

ELIGIBILITY:
Inclusion Criteria:

1. Baseline cTn measurement and at least one additional cTn measurement within 6 hours after initial measurement.
2. At least one 12-lead electrocardiogram

Exclusion Criteria:

1. Less than 18 years old
2. Pregnancy
3. Trauma
4. Decline to participate
5. Did not present through the ED
6. Transferred from an outside hospital or clinic.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consecutives patients (goal, 2000 patients over 4 months) presenting to the emergency department, in whom serial cTnI measurements are ordered on clinical indication at Hennepin Healthcare / Hennepin County Medical Center (Minneapolis, MN, USA) to rule-in and rule-out acute myocardial infarction.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Actual)
Dates: Start 2020-10-13 (Actual); Primary Completion 2021-10-13 (Actual); Study Completion 2024-10-13 (Actual)

PRIMARY OUTCOMES:
Incidence of acute myocardial infarction - Abbott hs-cTnI | Day 1
  Adjudicated diagnosis of acute myocardial injury using the Abbott hs-cTnI assay
Incidence of myocardial infarction - Roche Gen 5 cTnT | Day 1
  Adjudicated diagnosis of acute myocardial injury using the Roche Gen 5 cTnT assay
Incidence of myocardial infarction - Abbott contemporary cTnI | Day 1
  Adjudicated diagnosis of acute myocardial injury using the Abbott contemporary cTnT assay

SECONDARY OUTCOMES:
All-cause mortality | up to 180 days
  any death
Cardiac mortality | up to 180 days
  death due to cardiac reasons
Adjudicated index acute myocardial infarction according to 4th UDMI | on admission
  acute myocardial infarction, including sub-types following the Fourth Universal Definition of Myocardial Infarction
Number of participants that underwent revascularization | up to 180 days
  coronary artery bypass graft surgery or percutaneous coronary intervention
Safety Outcome - MACE | 30 days
  Major Adverse Cardiovascular Event - cardiac death, myocardial infarction, revascularization, congestive heart failure
Safety Outcome - MACE | 180 days
  Major Adverse Cardiovascular Event - cardiac death, myocardial infarction, revascularization, congestive heart failure

CONTACTS AND LOCATIONS:
Overall Officials: Fred S Apple, PhD, Principal Investigator — Hennepin Healthcare Research Institute
Locations (1):
- Hennepin Healthcare Research Institute / Hennepin County Medical Center, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Fabre-Estremera B, Smith SW, Sandoval Y, Schulz K, Okeson B, Cullen L, Apple FS. Rapid Rule-Out of Myocardial Infarction Using a Single High-Sensitivity Cardiac Troponin I Measurement Strategy at Presentation to the Emergency Department: The SAFETY Study. Clin Chem. 2023 Jun 1;69(6):627-636. doi: 10.1093/clinchem/hvad033. PMID 37022774